CLINICAL TRIAL: NCT00564148
Title: Intravitreal Injections With Avastin in Proliferative Retinopathies Related to the Production of VEGF Having Different Causes
Brief Title: Intravitreal Avastin in Proliferative Retinopathies
Acronym: SITE-App
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthalmological Association Edelweiss (Other)
Responsible Party: NARCISA IANOPOL, Ophthalmological Association Edelweiss
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVAST-ro-1; SITE-App
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-06

CONDITIONS: Retinal Neovascularization
Keywords: antiVEGF therapy
MeSH Terms: conditions — Retinal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A,1, II (Experimental)
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Avastin — 2,5 mg Avastin intravitreal injections every 4 weeks, 6 months consecutively
  Other Names: Bevacizumab

SUMMARY:
The study intends to assess the effect of Avastin injections in different proliferative retinopathies due to different causes

DETAILED DESCRIPTION:
Proliferative retinopathies due to different causes represent important causes for the visual acuity loss. Conventional treatments may sometimes improve the visual function, whereas other times, the visual acuity continue to decrease, in spite of all the medical, surgical or laser treatments.

Intravitreal injections with anti-VEGF agents (ex. Avastin for our trial) seem to be an important tool for certain difficult situations in which at the ocular fundus, out of different reasons (advanced age, diabetes mellitus, retinal veins occlusions, etc)new pathologic vessels appear, causing devastating changes in the posterior and anterior segment as well.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of a proliferative retinopathy (AGE RELATED MACULAR DEGENERATION,DIABETIC PROLIFERATIVE RETINOPATHY, etc)
* distance acuity < 0.5
* age > 20 years

Exclusion Criteria:

* noncooperative patients
* ocular infections / inflammations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The following parameters will be assessed in order to evaluate the Avastin effect: visual acuity, lesions's area at the ocular fundus | one year

SECONDARY OUTCOMES:
The intraocular pressure will be measured during the whole study in order to assess the possible side effects of Avastin injections | one year

CONTACTS AND LOCATIONS:
Overall Officials: NARCISA IANOPOL, researcher, Principal Investigator — Ophthalmological Association Edelweiss
Locations (1):
- Ochiul Diabetic, Iași, Romania